CLINICAL TRIAL: NCT05925946
Title: Effect of Low-Calorie Diet and Lifestyle Intervention on Reversal of Type 2 Diabetes Mellitus, Hepatic and Pancreatic Fat: A Two-year Randomized Control Trial in New Delhi, India
Brief Title: Effect of Low-Calorie Diet and Lifestyle Intervention on Reversal of T2DM
Acronym: CURE-DM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Foundation, India (Other)
Collaborators: Ministry of Science and Technology, India (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-1312
Record Dates: First submitted 2023-06-13; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus; PreDiabetes; Diet Habit
Keywords: Type 2 Diabetes, Low calorie diet, Asian Indians, hepatic fat, pancreatic fat
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Feeding Behavior; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 1. Phase1 (Partial diet replacement) (850 Kcal/day) (12-20 weeks)):
  2. Phase 2 (Gradual increase in calories) (20-28 weeks) (1100 Kcal/day):
  3. Phase 3 (Weight loss maintenance) (29-104 weeks) (up to 1200Kcal/day) :
  Interventions: Dietary Supplement: CURE-DM
- Control Group (No Intervention): Subjects will be given routine care for diabetes and obesity management with no change in medication. The meal plan for the control group will consist of 1400 Kcal/day achieved through small frequently distributed meals constituting around 15% of protein, 60% of carbohydrates and 25% of fat; with a menu resembling standard Indian dietary patterns and meal combinations.

INTERVENTIONS:
Dietary Supplement: CURE-DM — 1. This randomized controlled prospective trial will be of 2 years duration where 150 patients with T2DM from urban areas of Delhi will be screened.
  2. These subjects will be randomized into two groups by computer-generated randomization list using variable block size.
  3. Group A (n, 60, test group)will be received a low-calorie diet along with appropriate exercise counseling; and group B (n, 60, Control group) will be received balanced diet along with exercise advice.
  Arms: Intervention Group

SUMMARY:
An increase in body fat, even when within the normal BMI range is one of the essential drivers of T2DM in Asian Indians. In this context, the relationship between excess hepatic fat and pancreatic fat appears to be necessary. A low-calorie (high protein and low carb) vegetarian diet with appropriate exercise, in a protocol similar to the DiRECT study, may lead to weight loss, reversal of diabetes, and decrease in ectopic fat.

DETAILED DESCRIPTION:
Diabetes is one of the biggest global public health problems. India has 100 million people living with diabetes as per the 2023 data. Reversal of T2DM, the holy grail of diabetes management, was not deemed possible until recently. Primary care-led weight management for remission of type 2 diabetes (DiRECT) trial has been conducted in obese patients with T2DM patients for a period of 2 years in the UK. Research on the effect of dietary intervention would be necessary for Asian Indians since liver fat deposition is more severe than in white Caucasians. Although some nutritionists and physicians are replicating methods of DiRECT study in their patients, it is not clear if similar diets will work effectively in community-dwelling Asian Indians.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T2DM within the previous 3 years
* Age 20-65 years
* BMI >25-45kg/m2
* HbA1c> 6.5% at baseline (on current treatment, if any)

Exclusion criteria:

* Recent or screening HbA1c of 9% or higher
* Weight loss of >5 kg within the previous 6 months
* Significant cardiopulmonary
* Hepatic, or another endocrine disease
* Current participation in any other research drug study in the previous three months
* Past history of bariatric surgery Malignancy other than minor skin lesions and Possibility of pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Reversal of diabetes | 24 Months
  This randomized controlled prospective trial will be of 2 years duration with T2D. These subjects will be randomized into two groups, Group A (intervention group) will receive a professionally supported low-calorie diet along with appropriate exercise counselling; Group B (Control group) will be receiving encouragement to follow standard diet and exercise advice.

SECONDARY OUTCOMES:
Muscle strength | 24 Months
  Handgrip muscle strength by Jamar Dynamometer
Anthropometric assessment | 24 Months
  Weight, BMI, circumferences (waist, hip, mid-thigh, mid-arm and neck), skinfold thickness (biceps, triceps, sub scapular, supra-iliac, thigh, lateral thoracic and calf)
Hepatic and Pancreatic Fat | 24 Months
  Liver and pancreatic fat fraction (proton-density fat fraction-magnetic resonance imaging (PDFF-MRI) and thigh skeletal muscle area (by MRI).
Body fat | 24 Months
  Body fat will be done by Whole body dual-energy X-ray absorptiometry (DEXA scan
Insulin Resistance | 24 Months
  Surrogate markers of insulin sensitivity

IPD SHARING:
Plan to Share IPD: Undecided
This randomized controlled prospective trial will be of 2 years duration